CLINICAL TRIAL: NCT02229162
Title: Delayed Umbilical Cord Clamping For Term Infants: A Pilot Safety Trial During Cesarean Deliveries
Brief Title: Delayed Umbilical Cord Clamping - C-section Pilot
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 400656-4
Record Dates: First submitted 2014-07-22; First posted 2014-09-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2016-02

CONDITIONS: Cesarean Sections
Keywords: umbilical cord; cesarean section; Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 90 seconds DCC: the initial 15-20 subjects (15 enrolled subjects who complete study) will have cord clamped at 90 seconds. Then data will be analyzed and evaluated by DSMB
- Two minutes DCC: If Data Safety Monitoring Board (DSMB) concurs, DCC will then be practiced for 2 minutes for second group, which is the minimum amount of time recommended to be defined as DCC.

SUMMARY:
This is a pilot study of delayed cord clamping (DCC) at progressively longer intervals (90 to 120 seconds) during elective cesarean deliveries of term infants. The investigators hypothesize that the pilot trial of DCC in cesarean sections will demonstrate safety of this procedure for mothers and babies.

DETAILED DESCRIPTION:
Despite expert recommendations to delay clamping the cord for at least 2 minutes, early cord clamping remains a common obstetrical practice. The World Health Organization has noted that data on cesarean deliveries are more limited, particularly with respect to long-term effects in infants. Recently, the American College of Obstetrics and Gynecology also noted in a committee statement that " the ideal time for clamping of the umbilical cord in cesarean section vs. vaginal birth is a particularly important area for future research".

The objective of this study is to conduct a pilot trial of delayed cord clamping during cesarean deliveries to determine if progressively longer intervals of cord clamping are feasible and not related to poorer maternal and neonatal outcomes as compared to outcomes from historical controls. We will offer study entry for women planning elective cesarean delivery to collect prospective data on progressively longer intervals, analyzing outcomes for each time interval to ensure they are clinically acceptable, prior to extending the interval another 30 s. We anticipate approximately 20 women at each interval (90 and 120 sec) and will perform hemoglobin analysis on the infants specifically for this study. If intraoperative blood loss is clinically deemed excessive, or mother or baby are unstable, the cord will be clamped.

ELIGIBILITY:
Inclusion Criteria:Subjects that are pregnant (women 18 years of age and older) and scheduled for an elective C-section at ≥ 37 weeks gestation will be eligible for the study.

Exclusion Criteria:

Pregnant women that do not plan on having a C-section and individuals that are not pregnant. Pregnant women that are medically unstable, have poorly controlled diabetes mellitus, multiple gestations, anomalous fetuses and/or severe intrauterine growth retardation will be excluded. Adults unable to consent will not be included

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women 18 years of age or older that plan on having an elective Cesarean delivery of a term singleton infant.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
maternal estimated blood loss (EBL) | at delivery (approximately 1 hour duration)
  Excessive EBL will be assessed by three measures
  1. clinical assessment by anesthesia/obstetrics after surgery noting amount of blood suctioned and on drapes, to include weighing of drapes at > 800 mL
  2. difference between pre- and post-op hemoglobin levels of > 20% more than that in baseline data
  3. need for transfusion,

SECONDARY OUTCOMES:
neonatal hypothermia | at admission (within 30 minutes of birth)
  moderate or severe neonatal hypothermia (36.2 rectal or less)
newborn hemoglobin concentration and hematocrit | first day of life (0-24 h of age)
  mean hemoglobin concentration and incidence of polycythemia (hct >65 with symptoms, 70 without symptoms) and anemia (hgb <14.5 g/dL)

OTHER OUTCOMES:
phototherapy | < 14 days of age
  phototherapy for hyperbilirubinemia without evidence hemolysis during birth hospitalization or readmission during first 14 d of life
Neonatal intensive care (NICU) 'observation' or admission | birth hospitalization (first 72 h of age approximately)
  NICU 'observation' during transition or admission will be measured and reason for admission. respiratory symptoms are most of interest, but historical controls will only have data yes/no so we will look at overall nicu admissions also.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chantry, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chantry CJ, Blanton A, Tache V, Finta L, Tancredi D. Delayed cord clamping during elective cesarean deliveries: results of a pilot safety trial. Matern Health Neonatol Perinatol. 2018 Jul 4;4:16. doi: 10.1186/s40748-018-0083-3. eCollection 2018. PMID 29997897